CLINICAL TRIAL: NCT05247892
Title: Effectiveness of Ultrasound Versus Fluoroscopy Guided S1 Injections and Radiofrequency for the Management of Radicular Pain
Brief Title: Effectiveness of Ultrasound Versus Fluoroscopy Guided S1 Injections and Radiofrequency
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Diskapi Teaching and Research Hospital (Other)
Responsible Party: Principal Investigator, Selin Guven Kose, Medical Doctor, Diskapi Teaching and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 121/12
Record Dates: First submitted 2022-02-01; First posted 2022-02-21 (Actual); Last update posted 2022-11-02 (Actual); Status verified 2022-10

CONDITIONS: Pain, Chronic
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fluoroscopic-guided S1 Radiofrequency stimulation (Active Comparator)
  Interventions: Procedure: Fluoroscopic-guided S1 Radiofrequency stimulation
- Ultrasound-guided S1 Radiofrequency stimulation (Experimental)
  Interventions: Procedure: Ultrasound-guided S1 Radiofrequency stimulation

INTERVENTIONS:
Procedure: Ultrasound-guided S1 Radiofrequency stimulation — Pulsed radiofrequency stimulation of the S1 dorsal root ganglia under ultrasound-guidance
  Arms: Ultrasound-guided S1 Radiofrequency stimulation
Procedure: Fluoroscopic-guided S1 Radiofrequency stimulation — Pulsed radiofrequency stimulation of the S1 dorsal root ganglia under fluoroscopy-guidance
  Arms: Fluoroscopic-guided S1 Radiofrequency stimulation

SUMMARY:
The investigators aim to compare the effect of ultrasound versus floroscopy guided pulsed radiofrequency treatment of the lumbar dorsal root ganglion (DRG) of S1 in patients with a chronic lumbosacral radicular pain.

ELIGIBILITY:
Inclusion Criteria:

* Persistent pain score ≥ 4 on VAS, not responding to traditional treatments
* Radicular pain in lumbar region for 3 months or more,
* Pattern of radiation suggestive for S1 pathology

Exclusion Criteria:

* Patient refusal
* Coagulopathy
* Uncooperative patients
* Malignant disorder or currently under treatment for a malignant disorder
* Pregnancy
* Leg pain due to localized hip or knee pathology

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2022-10-10 (Actual); Study Completion 2022-10-20 (Actual)

PRIMARY OUTCOMES:
Pain scores | baseline to 6 months post-procedure
  Visual analog scale (VAS) for pain at the follow-up time periods. The visual analog scale is a numerical scale from 0 to 10; with 0 representing no pain and 10 representing the worst pain imaginable.

SECONDARY OUTCOMES:
Oswestry Disability Index (ODI) | baseline to 6 months post-procedure
  Mean Change from Baseline in functional disability scores based on Oswestry Disability Index. 0% to 20% indicate minimal disability, 21% to 40% indicate moderate disability, 41%-60% indicates severe disability, 61%-80% means crippled and 81%-100% indicates that the patient is either bed-bound or exaggerating his/her symptoms.
Patient satisfaction Questionnaire | baseline to 6 months post-procedure
  Satisfaction was measured on a 1 to 5 scale,Using score: 5-Excellent, 4-Very Good, 3-Good, 2-Fair, and 1-Poor

CONTACTS AND LOCATIONS:
Locations (1):
- Diskapi Yildirim Beyazit Training and Research Hospital, Ankara, Turkey (Türkiye)